CLINICAL TRIAL: NCT03342664
Title: MIND: A Prospective, Multicenter Study of Artemis a Minimally Invasive Neuro Evacuation Device, in the Removal of Intracerebral Hemorrhage
Brief Title: MIND: Artemis in the Removal of Intracerebral Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11899
Record Dates: First submitted 2017-10-18; First posted 2017-11-17 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Hemorrhage; Brain Hemorrhage; Cerebral Parenchymal Hemorrhage; Intracerebral Hemorrhage
Keywords: ICH; Stroke; Cerebral Hemorrhage; Intracranial Hemorrhage; Hemorrhage; Cerebrovascular Disorders; Brain bleed
MeSH Terms: conditions — Cerebral Hemorrhage; Intracranial Hemorrhages; Stroke; Hemorrhage; Cerebrovascular Disorders

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either minimally invasive hematoma evacuation with the Artemis Neuro Evacuation Device with medical management (MIS group) or best medical management alone (2:1) (MM).
Who Masked: Outcomes Assessor
Masking Description: 180 day mRS is blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Artemis + Medical Management (MIS) (Experimental): Minimally invasive hematoma evacuation with the Artemis Neuro Evacuation Device with medical management
  Interventions: Device: Artemis + Medical Management
- Best Medical Management Alone (MM) (Active Comparator): Best medical management alone per standard of care at treating institution
  Interventions: Other: Best Medical Management Alone (MM)

INTERVENTIONS:
Device: Artemis + Medical Management — Subject will receive best MM in addition to the MIS procedure with Artemis.
  Other Names: MIS + MM
  Arms: Artemis + Medical Management (MIS)
Other: Best Medical Management Alone (MM) — Subject will receive best MM for ICH as determined by stroke physician following AHA/ESO guidelines.
  Other Names: MM; Control
  Arms: Best Medical Management Alone (MM)

SUMMARY:
The primary objective of this multicenter randomized controlled study is to compare the safety and efficacy of minimally invasive hematoma evacuation with the Artemis Neuro Evacuation Device to best medical management for the treatment of intracerebral hemorrhage (ICH).

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥ 18 and ≤ 80
2. Supratentorial ICH of volume ≥ 20 and ≤ 80 cc (measured using A x B X C/2 method)
3. Hemostasis as confirmed by no arterial spot sign (may perform additional scan(s) every 6 hours to demonstrate hemostasis)
4. NIHSS ≥ 6
5. GCS ≥ 5 and ≤ 15
6. Historical mRS 0 or 1
7. Symptom onset < 24 hours prior to initial CT/MR
8. MIS must be initiated within 72 hours of ictus/bleed
9. SBP must be < 180 mmHg and controlled at this level for at least 6 hours

Exclusion Criteria:

1. Imaging

   1. "Arterial Spot Sign" identified on final CTA indicating expanding hemorrhage
   2. Hemorrhagic lesion such as a vascular malformation (cavernous malformation, AVM etc.), aneurysm, and/or neoplasm
   3. Hemorrhagic conversion of an underlying ischemic stroke
   4. Infratentorial hemorrhage
   5. Primary thalamic ICH (where the center of the hemorrhage emulates from the thalamus)
   6. Associated intra-ventricular hemorrhage requiring treatment for IVH-related mass effect or shift due to trapped ventricle (EVD for ICP management is allowed)
   7. Midbrain extension/involvement
   8. Absolute contraindication to CTA, conventional angiography and MRA
2. Coagulation Issues

   1. Absolute requirement for long-term anti-coagulation (e.g., mechanical valve replacement (bio-prostatic valve is permitted), high risk atrial fibrillation)
   2. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency
   3. Platelet count < 100 x 10^3 cells/mm3 or known platelet dysfunction
   4. INR > 1.4, elevated prothrombin time or activated partial thromboplastin time (aPTT), which cannot be corrected or otherwise accounted for (i.e., lupus anti-coagulant)
   5. Use of direct factor Xa inhibitors (e.g. apixaban, rivaroxaban, fondaparinux) within last 48 hours
3. Patient Factors

   1. Traumatic ICH
   2. High risk atrial fibrillation (e.g., mitral stenosis with atrial fibrillation) and/or symptomatic carotid stenosis
   3. Requirement for emergent surgical decompression or uncontrolled ICP after EVD
   4. Unable to obtain consent per Institution Review Board/Ethics Committee policy
   5. Pregnancy or positive pregnancy test (either serum or urine). Women of child-bearing potential must have a negative pregnancy test prior to enrollment
   6. Severe active infection requiring treatment (e.g. sepsis or purulent wound) at the time of enrollment
   7. Renal failure indicated by creatinine > 2 mg/dL or undergoing dialysis
   8. Any comorbid disease or condition expected to compromise survival or ability to complete follow-up assessments through 365 days
   9. Based on investigator's judgement, patient is unwilling or unable to comply with protocol follow up appointment schedule
   10. Active drug or alcohol use or dependence that, in the opinion of the site investigator would interfere with adherence to study requirements
   11. Currently participating in another interventional (drug, device, etc) clinical trial. Patients in observational, natural history, and/or epidemiological studies not involving intervention are eligible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-09-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (27):
  - Abrazo Central, Phoenix, Arizona
  - UCLA, Los Angeles, California
  - Mission Hospital, Mission Viejo, California
  - Swedish - HCA, Englewood, Colorado
  - Yale University, New Haven, Connecticut
  - Christiana Health, Newark, Delaware
  - George Washington, Washington D.C., District of Columbia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Loyola University Chicago, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - University of Mississippi, Jackson, Mississippi
  - University of Missouri, Columbia, Missouri
  - Atlantic Neuroscience Institute, Summit, New Jersey
  - Maimonides, Brooklyn, New York
  - Northwell Health, Manhasset, New York
  - Mount Sinai, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Novant Health, Charlotte, North Carolina
  - University Hospital Cleveland, Cleveland, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - MUSC, Charleston, South Carolina
  - Methodist University Hospital, Memphis, Tennessee
  - Valley Baptist Medical Center, Harlingen, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
- Uniklinikum Salzburg, Salzburg, Austria
- University of Alberta, Edmonton, Alberta, Canada
- Germany (4):
  - Universitätsklinikum Augsburg, Augsburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - München Klinik Bogenhausen, München

REFERENCES:
- [Derived] Arthur AS, Jahromi BS, Saphier PS, Nickele CM, Ryan RW, Vajkoczy P, Schirmer CM, Kellner CP, Matouk CC, Arias EJ, Ullman JS, Levitt MR, Hage ZA, Fiorella DJ; MIND Study Investigators and Collaborators. Minimally Invasive Surgery vs Medical Management Alone for Intracerebral Hemorrhage: The MIND Randomized Clinical Trial. JAMA Neurol. 2025 Nov 1;82(11):1113-1121. doi: 10.1001/jamaneurol.2025.3151. PMID 40892424

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Artemis + Medical Management (MIS) | Best Medical Management Alone (MM)
Started | 154 | 82
Completed | 139 | 70
Not Completed | 15 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Artemis + Medical Management (MIS) | Best Medical Management Alone (MM) | Total
Number analyzed (Participants) | 154 | 82 | 236
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (11.71) | 59.2 (12.33) | 59.4 (11.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 32 | 87
  Male | 99 | 50 | 149
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 9 | 31
  Not Hispanic or Latino | 115 | 61 | 176
  Unknown or Not Reported | 17 | 12 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 12 | 11 | 23
  Black or African American | 23 | 14 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 102 | 45 | 147
  More Than One Race | 2 | 0 | 2
  Other | 3 | 1 | 4
  Unknown | 1 | 4 | 5
  Not Reported | 10 | 7 | 17
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 1 | 3
  Austria | 0 | 1 | 1
  United States | 142 | 74 | 216
  Germany | 10 | 6 | 16
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.4 (8.21) | 30.9 (7.28) | 30.6 (7.88)

OUTCOME MEASURES:

1. Primary Outcome: Global Disability (Functional Outcome) Assessed Via the Ordinal Modified Rankin Score (mRS)
Description: Modified Rankin scale measures degree of disability or functional impairment on a scale of 0 (no symptoms) to 5 (severe disability), 6 (expired), where higher scores mean a worse outcome
Time Frame: 180 days
Population: As treated population
Measure: Count of Participants; unit: Participants
Groups:
- Artemis + Medical Management (MIS): Artemis + Medical Management (MIS) Minimally invasive hematoma evacuation with the Artemis Neuro Evacuation Device with medical management Artemis + Medical Management: Subject will receive best MM in addition to the MIS procedure with Artemis.
Arm/Group | Artemis + Medical Management (MIS) | Best Medical Management Alone (MM)
Number analyzed (Participants) | 154 | 82
Participants
  Missing mRS value | 32 | 20
  mRS 0 | 4 | 2
  mRS 1 | 5 | 1
  mRS 2 | 11 | 8
  mRS 3 | 28 | 14
  mRS 4 | 38 | 13
  mRS 5 | 14 | 10
  mRS 6 | 22 | 14
Statistical Analysis 1: Comparison: Artemis + Medical Management (MIS) vs Best Medical Management Alone (MM); Test type: Other; Odds Ratio (OR) = 1.03, 96% CI 2-sided [0.62 to 1.72] — Odds ratio of MIS over MM with value above 1 indicating a better outcome for MIS

2. Primary Outcome: Rate of Mortality
Time Frame: 30 days
Population: As treated population
Measure: Count of Participants; unit: Participants
Arm/Group | Artemis + Medical Management (MIS) | Best Medical Management Alone (MM)
Number analyzed (Participants) | 152 | 82
Participants | 11 | 8

3. Secondary Outcome: Functional Outcomes Measured Via Utility Weighted Modified Rankin Score (mRS)
Description: The utility-weighted modified Rankin Score (utility-weighted mRS) is a functional outcome measure that quantifies global disability. It is derived from the Ordinal Modified Rankin Scale (mRS), which assesses the degree of disability or functional impairment on a scale.
  The underlying Modified Rankin Scale categories range from 0 to 6, where:
  * 0 = No symptoms (best outcome)
  * 6 = Death (worst outcome)
  These categorical mRS values are converted to utility weights and the resulting the utility-weighted mRS produces a continuous score ranging from 0.00 to 1.00, where:
  * 0.00 represents the worst functional outcome (equivalent to severe disability or death)
  * 1.00 represents the best functional outcome (no symptoms and full independence)
  Higher scores indicate better functional outcomes. Lower scores indicate worse functional outcomes.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Artemis + Medical Management (MIS) | Best Medical Management Alone (MM)
Number analyzed (Participants) | 154 | 82
score on a scale | 0.41 (0.314) | 0.38 (0.318)

4. Secondary Outcome: Functional Outcomes Measured Via Modified Ordinal Rankin Score (mRS)
Description: as for outcome 1
Time Frame: 365 days
Population: As treated population
Measure: Count of Participants; unit: Participants
Groups:
- Artemis + Medical Management (MIS) All Participants All Participants: Artemis + Medical Management (MIS) Minimally invasive hematoma evacuation with the Artemis Neuro Evacuation Device with medical management Artemis + Medical Management: Subject will receive best MM in addition to the MIS procedure with Artemis.
Arm/Group | Artemis + Medical Management (MIS) All Participants All Participants | Best Medical Management Alone (MM)
Number analyzed (Participants) | 154 | 82
Participants
  Missing mRS value | 15 | 12
  mRS 0 | 4 | 0
  mRS 1 | 15 | 6
  mRS 2 | 11 | 15
  mRS 3 | 31 | 12
  mRS 4 | 45 | 14
  mRS 5 | 6 | 7
  mRS 6 | 27 | 16
Statistical Analysis 1: Comparison: Artemis + Medical Management (MIS) All Participants All Participants vs Best Medical Management Alone (MM); Test type: Other; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.64 to 1.79] — Odds ratio of MIS over MM with value above 1 indicating a better outcome for MIS

5. Secondary Outcome: Quality of Life Assessed Via Stroke Impact Scale
Description: The Stroke Impact Scale measures mobility and activities of daily living by assessing ability to perform specific physical tasks using a 5-point scale that ranges from 1 (could not do it at all) to 5 (not difficult at all). The individual scores are converted to a scale of 0 (no recovery) -100 (full recovery) to represent level of recovery, where a higher score means better outcome.
Time Frame: 180 and 365 days
Population: Numbers analyzed at 180 and 365 are dependent on data available from follow up visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Artemis + Medical Management (MIS) | Best Medical Management Alone (MM)
Number analyzed (Participants) | 154 | 82
score on a scale
  Mobility (180 days): number analyzed (Participants) | 91 | 45
  Mobility (180 days) | 54.3 (33.67) | 53.9 (34.19)
  Activities of Daily Living (180 days): number analyzed (Participants) | 91 | 45
  Activities of Daily Living (180 days) | 53.4 (31.89) | 53.8 (32.59)
  Mobility (365 days): number analyzed (Participants) | 91 | 41
  Mobility (365 days) | 55.0 (32.51) | 58.4 (33.99)
  Activities of Daily Living (365 days): number analyzed (Participants) | 91 | 41
  Activities of Daily Living (365 days) | 55.8 (30.66) | 56.2 (33.40)

6. Secondary Outcome: VAS Quality of Life Assessed Via EQ-5D-5L
Description: The EQ-5D-5L (EuroQol 5 Dimension 5 Level) is a self assessment on activities of daily living using a visual analog scale (VAS) where current health is rated on a scale of 0 to 100 where 0 is the worst imaginable health and 100 is the best imaginable health.
Time Frame: 180 and 365 days
Population: The number analyzed at 180 and 365 days are dependent on data available for participants completing visits.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Artemis + Medical Management (MIS) | Best Medical Management Alone (MM)
Number analyzed (Participants) | 154 | 82
score on a scale
  EQ-5D-5L-180 days: number analyzed (Participants) | 98 | 53
  EQ-5D-5L-180 days | 61.6 (23.41) | 62.4 (22.82)
  EQ-5D-5L-365 days: number analyzed (Participants) | 100 | 47
  EQ-5D-5L-365 days | 62.7 (22.42) | 66.0 (22.03)

7. Secondary Outcome: Length of Hospital Stay
Time Frame: Admission to hospital discharge (up to one year)
Population: All subjects
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Artemis + Medical Management (MIS) | Best Medical Management Alone (MM)
Number analyzed (Participants) | 140 | 77
days | 18.8 (17.81) | 20.6 (12.75)

8. Secondary Outcome: Length of ICU
Time Frame: # of days from admission (up to one year)
Population: All subjects
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Artemis + Medical Management (MIS) | Best Medical Management Alone (MM)
Number analyzed (Participants) | 140 | 77
days | 7.6 (6.51) | 9.2 (8.39)

9. Secondary Outcome: Length of Procedure
Time Frame: Time from initial sheath placement to final sheath removal
Population: all subjects (ITT), one participant was randomized to MM but received MIS treatment
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Artemis + Medical Management (MIS) | Best Medical Management Alone (MM)
Number analyzed (Participants) | 149 | 1
minutes | 41 (29.81) | 34 (NA) — There is only one participant in this group. Standard deviation is not available.

10. Secondary Outcome: Functional Outcomes Measured Via Modified Rankin Score (mRS) of ≤ 3
Description: (0 no symptoms - 3 moderate disability)
Time Frame: 180 days
Population: All subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Artemis + Medical Management (MIS) | Best Medical Management Alone (MM)
Number analyzed (Participants) | 138 | 76
Participants | 57 | 32

11. Secondary Outcome: Functional Outcomes Measured Via Modified Rankin Score (mRS) of ≤ 2
Description: mRS 0 no symptoms - 2 slight disability
Time Frame: 180 days
Population: All subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Artemis + Medical Management (MIS) | Best Medical Management Alone (MM)
Number analyzed (Participants) | 138 | 76
Participants | 26 | 14

ADVERSE EVENTS:
Time Frame: Within 365 days
Arm/Group | Artemis + Medical Management (MIS) | Best Medical Management Alone (MM)
All-Cause Mortality (participants affected / at risk) | 27/154 | 16/82
Serious Adverse Events (participants affected / at risk) | 89/154 | 60/82
Other Adverse Events (participants affected / at risk) | 107/154 | 56/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Artemis + Medical Management (MIS) (N=154) | Best Medical Management Alone (MM) (N=82)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiomegaly (Cardiac disorders) | 0 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 0
Visual impairment (Eye disorders) | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0
Chest pain (General disorders) | 1 | 2
Impaired healing (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0
Oedema peripheral (General disorders) | 0 | 0
Pain (General disorders) | 0 | 0
Pyrexia (General disorders) | 1 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Blister infected (Infections and infestations) | 1 | 0
Burn infection (Infections and infestations) | 0 | 0
COVID-19 (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Eye infection bacterial (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 0
Liver abscess (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 3
Parotitis (Infections and infestations) | 0 | 0
Pneumonia (Infections and infestations) | 4 | 7
Pneumonia escherichia (Infections and infestations) | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pneumonia streptococcal (Infections and infestations) | 0 | 0
Post procedural pneumonia (Infections and infestations) | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0
Pulmonary sepsis (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 4 | 9
Septic encephalopathy (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 3 | 0
Sputum purulent (Infections and infestations) | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0
Taeniasis (Infections and infestations) | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 2
Urosepsis (Infections and infestations) | 2 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 | 1
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Unintentional medical device removal (Injury, poisoning and procedural complications) | 0 | 2
Urethral injury (Injury, poisoning and procedural complications) | 0 | 0
Weaning failure (Injury, poisoning and procedural complications) | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0
Bacterial test positive (Investigations) | 0 | 0
Haemoglobin increased (Investigations) | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0
Liver function test increased (Investigations) | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0
Transaminases increased (Investigations) | 0 | 0
Troponin increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 0
Alcoholic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0
Cerebral salt-wasting syndrome (Metabolism and nutrition disorders) | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0
Brain midline shift (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 4 | 10
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 17 | 3
Cerebral infarction (Nervous system disorders) | 4 | 2
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Cytotoxic oedema (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0
Embolic cerebral infarction (Nervous system disorders) | 0 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0
External hydrocephalus (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 7 | 2
Headache (Nervous system disorders) | 0 | 0
Hemiparesis (Nervous system disorders) | 2 | 1
Hydrocephalus (Nervous system disorders) | 2 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0
IIIrd nerve paralysis (Nervous system disorders) | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 3 | 4
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0
Migraine (Nervous system disorders) | 1 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0
Paroxysmal sympathetic hyperactivity (Nervous system disorders) | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0
Seizure (Nervous system disorders) | 6 | 1
Somnolence (Nervous system disorders) | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 1
Stroke in evolution (Nervous system disorders) | 2 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 0
Subdural hygroma (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0
Mental status changes (Psychiatric disorders) | 2 | 0
Staring (Psychiatric disorders) | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 3
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Total (Skin and subcutaneous tissue disorders) | 2 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0
Subdural haematoma evacuation (Surgical and medical procedures) | 0 | 0
Tracheostomy (Surgical and medical procedures) | 0 | 0
Deep vein thrombosis (Vascular disorders) | 9 | 9
Haematoma (Vascular disorders) | 0 | 0
Hypertension (Vascular disorders) | 0 | 2
Hypertensive emergency (Vascular disorders) | 1 | 0
Hypertensive urgency (Vascular disorders) | 0 | 0
Hypotension (Vascular disorders) | 0 | 1
Poor venous access (Vascular disorders) | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Artemis + Medical Management (MIS) (N=154) | Best Medical Management Alone (MM) (N=82)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 6 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0
Diplopia (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 15 | 12
Enterocolitis (Gastrointestinal disorders) | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 13 | 6
Total (Hepatobiliary disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 1
Total (Immune system disorders) | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0
Total (Infections and infestations) | 41 | 20
Anal abscess (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Blister infected (Infections and infestations) | 0 | 0
Burn infection (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0
Eye infection bacterial (Infections and infestations) | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 16 | 7
Pneumonia escherichia (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Post procedural pneumonia (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 0
Sepsis (Infections and infestations) | 2 | 2
Septic encephalopathy (Infections and infestations) | 0 | 0
Septic shock (Infections and infestations) | 0 | 0
Sputum purulent (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Taeniasis (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 17 | 7
Urosepsis (Infections and infestations) | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 | 0
Haematuria traumatic (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0
Unintentional medical device removal (Injury, poisoning and procedural complications) | 0 | 1
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0
Weaning failure (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Bacterial test positive (Investigations) | 1 | 0
Haemoglobin increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
Troponin increased (Investigations) | 1 | 0
White blood cell count increased (Investigations) | 1 | 0
Alcoholic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Cerebral salt-wasting syndrome (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 4 | 6
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Brain midline shift (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 4 | 0
Cerebral infarction (Nervous system disorders) | 2 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Cytotoxic oedema (Nervous system disorders) | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 0
Encephalopathy (Nervous system disorders) | 3 | 0
Epilepsy (Nervous system disorders) | 0 | 1
External hydrocephalus (Nervous system disorders) | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 2 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0
Headache (Nervous system disorders) | 5 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 1
Intraventricular haemorrhage (Nervous system disorders) | 4 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 0
Muscle spasticity (Nervous system disorders) | 1 | 1
Neurological decompensation (Nervous system disorders) | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Paroxysmal sympathetic hyperactivity (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 12 | 7
Somnolence (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 0
Stroke in evolution (Nervous system disorders) | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0
Subdural hygroma (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0
Tremor (Nervous system disorders) | 2 | 0
Agitation (Psychiatric disorders) | 1 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 3 | 0
Delirium (Psychiatric disorders) | 5 | 0
Mental status changes (Psychiatric disorders) | 1 | 2
Staring (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 3
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0
Urinary retention (Renal and urinary disorders) | 8 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Respiratory tract oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Subdural haematoma evacuation (Surgical and medical procedures) | 0 | 1
Tracheostomy (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 5 | 4
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypertensive emergency (Vascular disorders) | 0 | 0
Hypertensive urgency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 3
Poor venous access (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 1
Thrombophlebitis superficial (Vascular disorders) | 5 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT03342664/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT03342664/SAP_001.pdf